CLINICAL TRIAL: NCT04330040
Title: A Prospective, Multicentre, Phase-IV Clinical Trial of Olaparib in Indian Patients With Platinum Sensitive Relapsed Ovarian Cancer Who Are in Complete or Partial Response Following Platinum Based Chemotherapy and Metastatic Breast Cancer With Germline BRCA1/2 Mutation
Brief Title: Prospective Multicentre Phase-IV Clinical Trial of Olaparib in Indian Patients With Ovarian and Metastatic Breast Cancer
Acronym: SOLI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0816R00025
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Breast Cancer
Keywords: Ovarian Cancer; Breast Cancer, Olaparib
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: A Prospective, Multicentre, Phase-IV Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Intervention: Drug: Olaparib
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Tablet

SUMMARY:
A Prospective, Multicentre, Phase-IV Clinical Trial of Olaparib in Indian Patients with Platinum Sensitive Relapsed Ovarian Cancer who are in Complete or Partial Response Following Platinum based Chemotherapy and Metastatic Breast Cancer with germline BRCA (BReast CAncer gene) 1/2 Mutation

DETAILED DESCRIPTION:
A Prospective, Multicentre, Phase-IV Clinical Trial of Olaparib in Indian Patients with Platinum Sensitive Relapsed Ovarian Cancer who are in Complete or Partial Response Following Platinum based Chemotherapy and Metastatic Breast Cancer with germline BRCA(BReast CAncer gene)1/2 Mutation As per recommendation from DCGI(Drug Controller general of of India), the current phase-IV study is planned with the aim to assess the safety in Indian subjects receiving olaparib as per the approved label indications in India in accordance with the requirements of the Health Authorities of India. This study attempts to descriptively elucidate the safety of Olaparib in Indian subjects receiving olaparib as per the Indian regulatory approved indications in India. The data obtained from the present study will help to understand the safety profile of olaparib in Indian patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures..
2. Female Subjects with ≥ 18 years of age
3. Subjects receiving olaparib for the following indications in ovarian cancer:

   for the maintenance treatment of adult subjects with recurrent epithelial ovarian, fallopian tube or primary peritoneal cancer, who are in a complete or partial response to platinum-based chemotherapy
4. Subjects receiving olaparib for the following indication in breast cancer:

in subjects with deleterious or suspected deleterious gBRCAm, HER2-negative metastatic breast cancer who have previously been treated with chemotherapy in the neoadjuvant, adjuvant or metastatic setting. Subjects with HR-positive breast cancer should have been treated with a prior endocrine therapy or be considered inappropriate for endocrine treatment

Exclusion Criteria:

1. Patients with either the history of hypersensitivity to excipients of the study drug or to drugs with a similar chemical structure or class to the study drug.
2. pregnant and/or lactating women.
3. Patients with a previously or currently diagnosed MDS/ AML or pneumonitis.
4. Patients who have not recovered sufficiently from prior surgery or anticancer treatment.
5. Patients who have known history of hepatitis B or hepatitis C
6. Patients with active infection such as TB.
7. Participation in another clinical study with a study drug administered in the last 3 months

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Bhubaneswar
  - Research Site, Chandigarh
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Guwahati
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, New Delhi
  - Research Site, Vellore

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816R00025&attachmentIdentifier=8803a976-d3b3-4269-9061-8c64c0adac18&fileName=d0816r00025-protocol-redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816R00025&attachmentIdentifier=00a5d0a0-5bf4-4d9b-a482-ea9e075eac26&fileName=d0816r00025-sap-redacted.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816R00025&attachmentIdentifier=b7184467-ff6a-425a-a6cf-16e0612c00e9&fileName=d0816r00025-synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were prescribed olaparib by an independent clinical judgement of investigator in his/her routine practice based on locally approved prescribing information were eligible for screening under this study.
Groups:
- Ovarian Cancer; Breast Cancer; Both Ovarian Cancer and Breast Cancer: Olaparib was administered orally at a dose of 300 mg (two 150-mg tablets) twice a day in all cohorts from Day 1 (Visit 2) to Day 182 (+/- 3 days; Visit 8).
Period: Overall Study
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian Cancer and Breast Cancer
Started | 163 | 38 | 1
Completed | 104 | 18 | 1
Not Completed | 59 | 20 | 0
Not completed — Other: Adverse event | 5 | 0 | 0
Not completed — Disease progression | 38 | 10 | 0
Not completed — Physician Decision | 5 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 2 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0
Not completed — Other: Increased QTc interval and clinical progression found | 0 | 1 | 0
Not completed — Other: Progressive disease (no confirming documents) | 0 | 1 | 0
Not completed — Other: Disease progression | 1 | 0 | 0
Not completed — Other: Due to anemia the investigator decided not to continue | 1 | 0 | 0
Not completed — Other: Due to disease progression and could not tolerate the dose | 1 | 0 | 0
Not completed — Enrolled and did not receive study drug (not included in Safety Analysis Set) | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian Cancer and Breast Cancer | Total
Number analyzed (Participants) | 163 | 38 | 1 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (8.78) | 44.3 (11.85) | 57.0 (NA) — Not evaluable - only one participant in this category | 51.5 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 38 | 1 | 202
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.204 (4.5366) | 24.699 (4.7282) | 21.210 (NA) — Only one participant in this category | 25.896 (4.6000)
Child Bearing Potential [Count of Participants; unit: Participants]
  Yes | 1 | 12 | 0 | 13
  No | 162 | 26 | 1 | 189
Stage/FIGO Stage of Cancer at Screening [Count of Participants; unit: Participants] — The higher the stage and grade of the cancer, the larger the tumor and the more it has spread. Cancers that are in higher stages have a worse prognosis.
  Participants
    Stage IA | 4 | 2 | 0 | 6
    Stage IB | 0 | 1 | 0 | 1
    Stage IC | 5 | 0 | 0 | 5
    Stage IIA | 1 | 3 | 0 | 4
    Stage IIB | 2 | 1 | 0 | 3
    Stage IIIA | 12 | 3 | 0 | 15
    Stage IIIB | 6 | 3 | 0 | 9
    Stage IIIC | 60 | 9 | 0 | 69
    Stage IVA | 42 | 10 | 1 | 53
    Stage IVB | 29 | 6 | 0 | 35
    Missing | 2 | 0 | 0 | 2
Previous Cancer Therapy [Count of Participants; unit: Participants]
  1 cancer therapy regimen | 2 | 8 | 0 | 10
  2 cancer therapy regimens | 55 | 10 | 1 | 66
  More than 2 cancer therapy regimens | 106 | 19 | 0 | 125
  No | 0 | 1 | 0 | 1
WHO Performance Status [Count of Participants; unit: Participants] — WHO = World Health Organization
  Participants
    Normal activity | 157 | 38 | 1 | 196
    Restricted activity | 6 | 0 | 0 | 6
    In bed less than or equal to 50% of the time | 0 | 0 | 0 | 0
    In bed more than 50% of the time | 0 | 0 | 0 | 0
    100% bedridden | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Haematology: Basophils Absolute Count, Eosinophils Absolute Count, Leucocytes WBC, Lymphocytes Absolute Count, Monocytes Absolute Count, Neutrophils Absolute Count, and Platelets Parameters
Description: The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib. Comparison between the cohorts was not the objective for the study. The hematology data were analyzed as above normal/normal/below normal and are presented as end of treatment status for the overall population .
  EOT = end of treatment
Time Frame: Baseline to EOT (approximately 6 months)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Groups:
- Ovarian; Breast Cancer; Both Ovarian and Breast Cancer: Olaparib was administered orally at a dose of 300 mg (two 150-mg tablets) twice a day in all cohorts from Day 1 (Visit 2) to Day 182 (+/- 3 days; Visit 8).
- Cancer Type: Overall: All participants included in this analysis
Arm/Group | Ovarian | Breast Cancer | Both Ovarian and Breast Cancer | Cancer Type: Overall
Number analyzed (Participants) | 161 | 38 | 1 | 200
Participants
  Basophils Absolute Count: EOT Above Normal | 0 | 0 | 0 | 0
  Basophils Absolute Count: EOT Normal | 72 | 12 | 1 | 85
  Basophils Absolute Count: EOT Below Normal | 41 | 10 | 0 | 51
  Basophils Absolute Count: EOT Missing | 48 | 16 | 0 | 64
  Eosinophils Absolute Count: EOT Above Normal | 2 | 0 | 0 | 2
  Eosinophils Absolute Count: EOT Normal | 90 | 20 | 1 | 111
  Eosinophils Absolute Count: EOT Below Normal | 21 | 3 | 0 | 24
  Eosinophils Absolute Count: EOT Missing | 48 | 15 | 0 | 63
  Leucocytes WBC: EOT Above Normal | 2 | 1 | 0 | 3
  Leucocytes WBC: EOT Normal | 101 | 17 | 1 | 119
  Leucocytes WBC: EOT Below Normal | 27 | 8 | 0 | 35
  Leucocytes WBC: EOT Missing | 31 | 12 | 0 | 43
  Lymphocytes Absolute Count: EOT Above Normal | 0 | 0 | 0 | 0
  Lymphocytes Absolute Count: EOT Normal | 79 | 10 | 0 | 89
  Lymphocytes Absolute Count: EOT Below Normal | 51 | 16 | 1 | 68
  Lymphocytes Absolute Count: EOT Missing | 31 | 12 | 0 | 43
  Monocytes Absolute Count: EOT Above Normal | 3 | 1 | 0 | 4
  Monocytes Absolute Count: EOT Normal | 84 | 14 | 1 | 99
  Monocytes Absolute Count: EOT Below Normal | 26 | 8 | 0 | 34
  Monocytes Absolute Count: EOT Missing | 48 | 15 | 0 | 63
  Neutrophils Absolute Count: EOT Above Normal | 2 | 1 | 0 | 3
  Neutrophils Absolute Count: EOT Normal | 107 | 19 | 1 | 127
  Neutrophils Absolute Count: EOT Below Normal | 21 | 6 | 0 | 27
  Neutrophils Absolute Count: EOT Missing | 31 | 12 | 0 | 43
  Platelets: EOT Above Normal | 18 | 6 | 1 | 25
  Platelets: EOT Normal | 69 | 13 | 0 | 82
  Platelets: EOT Below Normal | 43 | 7 | 0 | 50
  Platelets: EOT Missing | 31 | 12 | 0 | 43

2. Primary Outcome: Haematology: Haemoglobin Parameters
Description: The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib. The haemoglobin parameter data were analyzed as above normal/normal/below normal and are presented as end of treatment status for the overall population .
  EOT = end of treatment
Time Frame: Baseline to EOT (approximately 6 months)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian and Breast Cancer | Cancer Type: Overall
Number analyzed (Participants) | 161 | 38 | 1 | 200
Participants
  EOT Above Normal | 0 | 0 | 0 | 0
  EOT Normal | 15 | 5 | 0 | 20
  EOT Below Normal | 115 | 21 | 1 | 137
  EOT Missing | 31 | 12 | 0 | 43

3. Primary Outcome: Number of Participants Who Experienced a Shift in Hematology Parameters to Results Classified as Below Normal at EOT
Description: The number of participants who experienced hematology results classified as normal at Baseline which shifted to below normal at the End of Treatment visit are presented.
  The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib.
  EOT = end of treatment
Time Frame: Baseline to EOT (approximately 6 months)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian and Breast Cancer | Cancer Type: Overall
Number analyzed (Participants) | 161 | 38 | 1 | 200
Participants
  Basophils Absolute Count | 13 | 5 | 0 | 18
  Eosinophils Absolute Count | 8 | 2 | 0 | 10
  Leucocytes WBC | 17 | 6 | 0 | 23
  Lymphocytes Absolute Count | 20 | 8 | 1 | 29
  Monocytes Absolute Count | 21 | 6 | 0 | 27
  Neutrophils Absolute Count | 9 | 5 | 0 | 14
  Platelets | 23 | 4 | 0 | 27

4. Primary Outcome: Number of Participants Who Experienced a Shift in Hemoglobin Parameters to Results Classified as Below Normal at EOT
Description: The number of participants who experienced hemoglobin results classified as normal at Baseline which shifted to below normal at the End of Treatment visit are presented..
  The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib.
  EOT = end of treatment
Time Frame: Baseline to EOT (approximately 6 months)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian and Breast Cancer | Cancer Type: Overall
Number analyzed (Participants) | 161 | 38 | 1 | 200
Participants | 17 | 11 | 0 | 28

5. Primary Outcome: Number of Participants With Remarkable Changes in Clinical Chemistry Values Over Time as Assessed by Investigator
Description: The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib.
  Remarkable changes were assessed by the investigator.
  EOT = end of treatment
Time Frame: Baseline to EOT (approximately 6 months)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian and Breast Cancer
Number analyzed (Participants) | 161 | 38 | 1
Participants | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Remarkable Changes in Physical Examination Over Time as Assessed by Investigator
Description: Abnormal clinically significant results at Baseline and EOT are presented.
  The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib.
Time Frame: Baseline to EOT (approximately 6 months)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian Cancer and Breast Cancer
Number analyzed (Participants) | 161 | 38 | 1
Participants
  Abnormal Clinically Significant result at Baseline: Physical Examination Status | 0 | 0 | 0
  Abnormal Clinically Significant result at Baseline: General Appearance | 0 | 0 | 0
  Abnormal Clinically Significant result at Baseline: Respiratory | 0 | 0 | 0
  Abnormal Clinically Significant result at Baseline: Cardiovascular | 0 | 0 | 0
  Abnormal Clinically Significant result at Baseline: Abdomen | 0 | 0 | 0
  Abnormal Clinically Significant result at Baseline: Lymph Nodes | 0 | 0 | 0
  Abnormal Clinically Significant result at Baseline: Musculoskeletal system | 0 | 1 | 0
  Abnormal Clinically Significant result at Baseline: No response | 161 | 37 | 1
  Abnormal Clinically Significant result at End of Treatment: Physical Examination Status | 2 | 1 | 0
  Abnormal Clinically Significant result at End of Treatment: General Appearance | 0 | 0 | 0
  Abnormal Clinically Significant result at End of Treatment: Respiratory | 1 | 1 | 0
  Abnormal Clinically Significant result at End of Treatment: Cardiovascular | 0 | 0 | 0
  Abnormal Clinically Significant result at End of Treatment: Abdomen | 1 | 0 | 0
  Abnormal Clinically Significant result at End of Treatment: Lymph Nodes | 0 | 1 | 0
  Abnormal Clinically Significant result at End of Treatment: Musculoskeletal system | 0 | 0 | 0
  Abnormal Clinically Significant result at End of Treatment: No response | 157 | 35 | 1

7. Primary Outcome: Number of Participants With Remarkable Changes in Vital Signs Over Time as Assessed by Investigator
Description: as for outcome 5
Time Frame: Baseline to EOT (approximately 6 months)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian Cancer and Breast Cancer
Number analyzed (Participants) | 161 | 38 | 1
Participants | 0 | 0 | 0

8. Primary Outcome: WHO Performance Status
Description: The objective of this Phase 4 study was to assess the overall safety of Olaparib in participants with ovarian or breast cancer who were prescribed the drug in routine clinical practice based on locally approved prescribing information. The number of participants with ovarian or breast cancer planned to receive Olaparib was not predetermined and was dependent on patients in routine clinical practice eligible to receive Olaparib.
Time Frame: Baseline and End of study visit (200 days)
Population: The safety analysis set included all participants who received the study drug (200 overall).
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian and Breast Cancer | Cancer Type: Overall
Number analyzed (Participants) | 161 | 38 | 1 | 200
Participants
  Baseline: Normal activity | 155 | 38 | 1 | 194
  Baseline: Restricted activity | 6 | 0 | 0 | 6
  Baseline: In bed less than or equal to 50% of the time | 0 | 0 | 0 | 0
  End of Study: number analyzed (Participants) | 100 | 13 | 0 | 113
  End of Study: Normal activity | 92 | 12 | 0 | 104
  End of Study: Restricted activity | 7 | 1 | 0 | 8
  End of Study: In bed less than or equal to 50% of the time | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: Events with start date on or after the date of first dose of study treatment until 28 days after last dose of study treatment. Adverse events that were a consequence of a pre-existing condition that worsened later during the treatment phase (ie, events having start date before the date of first dose of study treatment and have worsened in severity while on study treatment) were termed as 'Treatment-emergent'.
  Adverse events for the Safety Analysis Set are presented.
Arm/Group | Ovarian Cancer | Breast Cancer | Both Ovarian Cancer and Breast Cancer
All-Cause Mortality (participants affected / at risk) | 3/161 | 3/38 | 0/1
Serious Adverse Events (participants affected / at risk) | 24/161 | 7/38 | 1/1
Other Adverse Events (participants affected / at risk) | 148/161 | 30/38 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovarian Cancer (N=161) | Breast Cancer (N=38) | Both Ovarian Cancer and Breast Cancer (N=1)
Anaemia (Blood and lymphatic system disorders) | 12 (14) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Aspiration pleural cavity (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ovarian Cancer (N=161) | Breast Cancer (N=38) | Both Ovarian Cancer and Breast Cancer (N=1)
Anaemia (Blood and lymphatic system disorders) | 82 | 14 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 35 | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 18 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 13 | 1 | 0
Nausea (Gastrointestinal disorders) | 33 | 3 | 0
Vomiting (Gastrointestinal disorders) | 27 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 14 | 1 | 0
Constipation (Gastrointestinal disorders) | 10 | 4 | 0
Fatigue (General disorders) | 25 | 3 | 0
Asthenia (General disorders) | 13 | 3 | 1
Pyrexia (General disorders) | 16 | 2 | 0
COVID-19 (Infections and infestations) | 8 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 18 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 3 | 0
Headache (Nervous system disorders) | 9 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2019-10-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04330040/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04330040/SAP_001.pdf